CLINICAL TRIAL: NCT05292651
Title: OPtimal stEnt Deployment stRategy oF Contemporary sTents
Acronym: PERFECTPSP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Schweitzer Hospital (Other)
Responsible Party: Principal Investigator, Dr. Rohit M. Oemrawsingh, Principal Investigator, Albert Schweitzer Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PERFECT 001
Record Dates: First submitted 2021-12-02; First posted 2022-03-23 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: single-center, prospective, single blinded randomized clinical trial
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PSP technique (Experimental): The definitions of the PSP technique are:
  * Predilatation is mandatory with a balloon diameter equal to or maximally 0.5 mm less than the distal reference vessel diameter. We hypothesize that this lesion preparation and fracture of the calcium may result in better stent apposition, less recoil and higher minimal stent area (MSA) Also see endpoints.
  * The DES should be deployed at 2 atm. above the nominal pressure. This relatively low stent deployment pressure may prevent stent edge dissections.
  * The postdilatation is mandatory with a shorter length and (at least 0.25mm) larger diameter non-compliant balloon at 16 atm. The apposition, minimal stent area (MSA) and recoil may improve with this large, high pressure postdilatation. The slightly shorter balloon can prevent edge dissections.
  Interventions: Procedure: PCI
- Direct Stenting (Active Comparator): • The DES is directly placed without any lesion preparation and deployed at a pressure at the discretion of the operator. Ideally a pressure would be achieved in which angiographic expansion of the DES is complete (without significant dog-boning)
  Interventions: Procedure: PCI

INTERVENTIONS:
Procedure: PCI — percutaneous coronary intervention

SUMMARY:
The primary objective is to evaluate whether a standard pre- and postdilatation (PSP strategy) of the modern DES results in a more optimal stent implantation compared to DS as evaluated by OCT in patients with stable coronary artery disease. The secondary clinical objective is to evaluate clinical cardiovascular outcomes in patients with stable coronary artery disease treated with the PSP strategy.

DETAILED DESCRIPTION:
Rationale: Historically, when coronary stents were initially introduced, the standard and mandatory treatment of a significant stenosis was with pre-dilation prior to stent placement. In the 2000s, several studies found no significant difference in clinical outcome between the two different stent implantation techniques: direct stenting (DS) versus the conventional stenting after pre-dilation (CS). Consequently, the stent implantation technique has become "unprotocolarised", i.e. each operator has their own, individual set of reasons for applying or avoiding pre- and post-dilation in specific conditions. However, these trials do not apply to the current/modern clinical practice of coronary stenting. The current patient population undergoing percutaneous coronary intervention (PCI) cannot be compared to the population that was treated in the early 2000s. The same applies for stent design. Stents have undergone several major transformations in the last 20 years. Furthermore, the events rates after PCI have significantly decreased within the last decades due to better stent design and improved background pharmacological therapy.

Imaging studies have revealed that an optimal stent result is not achieved in a high percentage of stent implantations. Post-hoc studies have demonstrated that the optimization of the implantation technique could reduce adverse cardiac events over time. As a result of these findings, the PSP concept: Pre-dilation, Sizing and Post-dilation was introduced. Whether routine pre- and postdilatation compared to DS also results in optimal stent implantation in contemporary drug-eluting stents (DES) has not been investigated and, hence is currently unknown.

Objective: The primary objective is to evaluate whether a standard pre- and postdilatation (PSP strategy) of the modern DES results in a more optimal stent implantation compared to DS as evaluated by OCT in patients with stable coronary artery disease. The secondary clinical objective is to evaluate clinical cardiovascular outcomes in patients with stable coronary artery disease treated with the PSP strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Stable angina patients or acute coronary syndrome patients with bystander stable coronary artery disease
2. With one or more significant epicardial stenosis in native coronary arteries suitable for direct stenting, according to the judgement of treating operator.

   The use of fractional flow reserve (FFR) or resting indices like iFR and RFR to assess lesion severity is encouraged.
3. Subject must be at least 18 years of age
4. Written consent to participate in the study

Exclusion Criteria:

1. Lesions not suitable for direct stenting, like (sub)-total stenosis, severely calcified lesions
2. Culprit lesions of acute coronary syndrome cannot be randomized to the trial. After successful treatment of the ACS culprit lesion, patients however can be randomized in the trial in case of remaining stable non-culprit lesions that thought to be stented directly of during a staged procedure.
3. Lesions not suitable for OCT catheter delivery and imaging, e.g. left main or ostial right coronary artery stenosis, lesions in coronary bypass grafts or tortuous anatomy
4. Treatment for in-stent restenosis
5. Bifurcation lesions in which a two-stent technique or a proximal postdilatation is planned.
6. Treatment of coronary artery bypass grafts
7. Creatine Clearance ≤ 30 ml/min/1.73 m2 (as calculated by MDRD formula for estimated GFR)
8. Known hypersensitivity or allergy for cobalt chromium
9. Known comorbidity associated with a life expectancy < 1 year
10. Unable to understand and follow study-related instructions or unable to comply with study protocol

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Suboptimal stent results which is defined as a composite of major stent underexpansion and major edge dissection measured by OCT at lesion level directly after completion of the stent implantation according to the protocol | During procedure
  Stent malapposition (categorical variable) is defined as:
  * Unacceptable stent expansion: The minimal stent area (MSA) of the proximal segment is <90% of the proximal lumen area, and/or the MSA of the distal segment is <90% of the distal reference lumen area on OCT OR
  * Presence of incompletely apposed stent struts on OCT more than 3mm long (defined as stent struts clearly separated from the vessel wall (lumen border/plaque border) without any tissue behind the struts with a distance from the adjacent intima of ≥0.2 mm and not associated with any side branch: i.e. the Prati criterium)
  Edge dissections (categorical variable) will be presented as:
  • Dissections on OCT of ≥60 degrees of the circumference of the vessel at the site of dissection and ≥3 mm in length

SECONDARY OUTCOMES:
Minimal stent area (MSA) (mm^2) | During procedure
Acute recoil (percent) | During procedure
  assessed on coronary angiography
Stent malapposition (percent) | During procedure
  defined as frequency of incompletely apposed stent struts (defined as stent struts clearly separated from the vessel wall (lumen border/plaque surface) without any tissue behind the struts with a distance from the adjacent intima of ≥0.2 mm and not associated with any side branch).
Mean stent expansion (percent): | During procedure
  mean stent area (stent volume/analysed stent length) divided by the average of proximal and distal reference lumen areas x 100
Intra-stent plaque protrusion and thrombus | During procedure
  defined as any intraluminal mass protruding at least 0.2 mm within the luminal edge of a stent strut
Post OCT stent result optimalization (percent) | During procedure
  composite of additional post-dilation and/or stent placements after OCT
MACE | 1-,3- and 5-year follow-up
  a composite of time- to-first event rate of cardiac death, target vessel MI, ischemia-driven target vessel revascularization (TVR)
Target Lesion Failure (TLF) | 1-,3- and 5-year follow-up
  defined as cardiac death, target vessel- myocardial infarction and clinically indicated target lesion revascularization)
Target Vessel Failure (TVF) | 1-,3- and 5-year follow-up
  defined as cardiac death, target vessel- myocardial infarction and clinically indicated target vessel revascularization
All cause mortality | 1-,3- and 5-year follow-up
Stent Thrombosis | 1-,3- and 5-year follow-up
  definite or probable; Academic Research Consortium (ARC) definition
Cost-effectiveness analysis | 1-,3- and 5-year follow-up
  total number of stent, balloons, wires and repeat hospitalizations due to MACE

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Oemrawsingh, MD, PhD, Principal Investigator — Albert Schweitzer Hospital
Locations (1):
- Albert Schweitzer hospital, Dordrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No